CLINICAL TRIAL: NCT05042284
Title: Effect of Non-enteric Coated Enzymes Substitution on Pain in Patients With Chronic Pancreatitis: a Double -Blinded Placebo Controlled Randomized Trial (NE-PERT Trial)
Brief Title: Effect of Non-enteric Coated Enzymes Substitution on Pain in Patients With Chronic Pancreatitis
Acronym: NE-PERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupjyoti Talukdar, Director, Pancreatology; Head, Pancreas Research Group and Division of Gut Microbiome Research, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NE PERT 1
Record Dates: First submitted 2021-08-20; First posted 2021-09-13 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pancreatitis; Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NE PERT (Experimental): Non-enteric coated pancreatic enzyme capsules containing 30,000U of protease will be provided three times a day along with food (breakfast, lunch and dinner)
  Interventions: Drug: Non-enteric coated pancreatic enzyme preparation
- Placebo (Placebo Comparator): Similar appearing glucose capsules will be provided three times a day along with food (breakfast, lunch and dinner)
  Interventions: Drug: Non-enteric coated pancreatic enzyme preparation

INTERVENTIONS:
Drug: Non-enteric coated pancreatic enzyme preparation — The patients will be given a non-enteric coated pancreatic enzyme capsule containing 30000 U of protease thrice daily along with meals for 3 months.
  Other Names: Placebo

SUMMARY:
Pain in CP entails several independent yet overlapping mechanisms including oxidative stress-mediated parenchymal inflammation, pancreatic and central neuropathy and neuroplasticity. Medical modalities for long-term pain management includes antioxidants and neuromodulators. Pancreatic enzymes are also invariably used for pain management. CP with ductal obstruction and pain is treated with either endotherapy or drainage surgery. However, it has been observed that a substantially increasing proportion of patients experience pain recurrence as the duration of follow-up after endotherapy or surgery gets longer.

Neural and dietary (proteins) stimuli activate CCK receptors in D1 & D2 which gives a positive feedback signal for pancreatic secretion. Once enzyme secretion starts, due to ductal and interstitial/tissue hypertension, nociception begins that results in pain. Blockade of the duodenal CCK receptors could inhibit the positive feedback loop, thereby reducing pancreatic secretion and resulting pain. Currently available enteric coated enzyme supplements are released throughout the small bowel and therefore may not be released sufficiently in the duodenum to effectively suppress the feedback loops. High doses of proteases (~25k-30k) would be required to block the receptors, while most of the currently available preparations have higher lipase but not proteases.

This led to the investigators' hypothesis that negative feedback of CCK by non enteric coated pancreatic enzymes could ameliorate pain in a more effective manner by NE-PERT.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is a fibro-inflammatory disorder of the pancreas characterized by progressive and irreversible damage. It manifests with abdominal pain and/or exocrine or endocrine insufficiency. Recurrent abdominal pain is the dominant clinical hallmark that mandates aggressive management. Pain in CP entails several independent yet overlapping mechanisms including oxidative stress-mediated parenchymal inflammation, pancreatic and central neuropathy and neuroplasticity.

Medical modalities for long-term pain management includes antioxidants and neuromodulators. Pancreatic enzymes are also invariably used for pain management. CP with ductal obstruction and pain is treated with either endotherapy or drainage surgery. However, it has been observed that a substantially increasing proportion of patients experience pain recurrence as the duration of follow-up after endotherapy or surgery gets longer.

It has been postulated that neural and dietary (proteins) stimuli activate CCK receptors in D1 & D2 which gives a positive feedback signal for pancreatic secretion. Once enzyme secretion from the pancreas begins, due to ductal and interstitial/tissue hypertension, nociception is initiated that results in pain. On this premise, the investigators hypothesized that blocking the duodenal CCK receptors could inhibit the positive feedback loop, thereby reducing pancreatic secretion and resulting pain.

Earlier meta-analyses that evaluated the effect of pancreatic enzyme supplementation on pain reported that there were no overall benefits in pain management. All but two of those studies used enteric coated enzyme. Currently available enteric coated enzyme supplements are released throughout the small bowel and therefore may not be released sufficiently in the duodenum to effectively suppress the feedback loops. High doses of proteases (~25k-30k) would be required to block the receptors, while most of the currently available preparations have higher lipase but not proteases. However, on subgroup analyses in the aforementioned meta-analyses, pain reduction was observed in the two studies that used non-enteric coated preparations. These studies were done several years earlier, had a small sample size, and had a cross over design. This formed that rationale of the investigators' current study to test the hypothesis using a statistically valid design with a higher sample size that would allow subgroup analyses, adjust for alternative pain mechanisms, and achieve a better effect size.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis of at least 3 years
* At least 3 episodes of pain in the past 3 months
* Pain score of at least 3 on VAS (0-10)
* Age 18-60yrs
* Both genders

Exclusion Criteria:

* Acute pancreatitis episode at the time of enrolment.
* Pancreatic cancer.
* Other chronic painful conditions.
* Active substance use (alcohol, smoking, smokeless tobacco, illicit drugs).
* Pregnancy and lactation.
* Inability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in pain score 1 | 3 months
  Visual analogue score will be used. Score ranges from 0-10, 10 indicating most severe.
Change in pain score 2 | 3 months
  Izbicki pain score will be used. Score ranges from 0-100, 100 indicating most severe.

SECONDARY OUTCOMES:
Change in pain score 1 | 6 months
  Visual analogue score will be used. Score ranges from 0-10, 10 indicating most severe.
Change in pain score 2 | 6 months
  Izbicki pain score will be used. Score ranges from 0-100, 100 indicating most severe.
Change in number of painful days | 3 months
  Number of days when the patient experienced pain
Change in number of painful days | 6 months
  Number of days when the patient experienced pain
Change in quality of life | 3 months
  Will be measured using the EORTC QLQ c30 with PAN28 tool. Score ranges from 0 to 100. 0 indicates worst for function scales, while 100 indicates worst for symptom scales.
Change in quality of life | 6 months
  Will be measured using the EORTC QLQ c30 with PAN28 tool. Score ranges from 0 to 100. 0 indicates worst for function scales, while 100 indicates worst for symptom scales.
Change in analgesic requirement | 3 months
  Number of analgesic tablets required will be recorded
Change in analgesic requirement | 6 months
  Number of analgesic tablets required will be recorded
Change in the number of hospitalization | 3 months
  Number of hospital admissions and days in hospital will be recorded
Change in the number of hospitalization | 6 months
  Number of hospital admissions and days in hospital will be recorded

OTHER OUTCOMES:
Change in Quantitative sensory testing parameters (pin prick) [First follow-up] | 3 months
  Pin prick sensation (0-10; 10 indicates maximum)
Change in Quantitative sensory testing parameters (pin prick) [Second follow-up] | 6 months
  Pin prick sensation (0-10; 10 indicates maximum);
Change in Quantitative sensory testing parameters (cold tolerance) [First follow-up] | 3 months
  Cold tolerance (0-10 VAS every 10secs for 2 mins.; 10 indicates severe)
Change in Quantitative sensory testing parameters (cold tolerance) [Second follow-up] | 6 months
  Cold tolerance (0-10 VAS every 10secs for 2 mins.; 10 indicates severe)
Change in pain DETECT score [First follow-up] | 3 months
  The painDETECT questionnaire will be used. Range is 0-38, 38 indicates most severe neuropathic pain.
Change in pain DETECT score [Second follow-up] | 6 months
  The painDETECT questionnaire will be used. Range is 0-38, 38 indicates most severe neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rupjyoti Talukdar, MD, AGAF, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After 6 months of data publication, on reasonable request.